CLINICAL TRIAL: NCT03538496
Title: Erector Spinae Plane Block Versus Thoracic Paravertebral Block on Postoperative Pain for Video Assisted Thoracoscopic Surgery
Brief Title: Comparison of Erector Spinae Plane Block With Thoracic Paravertebral Block for Video Assisted Thoracoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ali Ahiskalioglu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AUTF ANESTHESIA5
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound guided erector spinae plane block (Active Comparator): ultrasound guided erector spinae plane block with 20 ml %0.25 bupivacaine
  Interventions: Drug: Bupivacaine Hcl 0.25% Inj
- ultrasound guided paravertebral block (Active Comparator): ultrasound guided paravertebral block with 20 ml %0.25 bupivacaine
  Interventions: Drug: Bupivacaine Hcl 0.25% Inj

INTERVENTIONS:
Drug: Bupivacaine Hcl 0.25% Inj — Single shot 20 ml 0.25 bupivacaine

SUMMARY:
Erector Spinae Plane Block (ESPB) is a newly described and effective interfascial plane block for thoracic and abdominal surgery. It was first described by Forero et al. in 2016, effectiveness being reported in four cases. The paravertebral block has been successfully used in various surgical patient groups for purposes of anesthesia or postoperative pain management such as thoracotomy, breast surgery and abdominal surgery. The aim of this study is to compare the analgesic effects of erector spinae plane block and paravertebral block in patients undergoing video assisted thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-III patients
* Undergoing video assisted thoracoscopic surgery

Exclusion Criteria:

* chronic pain
* bleeding disorders
* renal or hepatic insufficiency
* patients on chronic non-steroidal anti-inflammatory medications
* emergency cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | First 24 hours
  First 24 hours total fentanyl consumption with patient controlled analgesia

SECONDARY OUTCOMES:
Visual analog pain score | postoperative 0-24 hours
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain)
Block performing time | First hour
  The block time was defined as the period between the insertion of the needle and termination of local anesthetic administration

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No